CLINICAL TRIAL: NCT05877443
Title: Barotrauma in Adults With Critical COVID-19
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sandra Jonmarker, Consultant in intensive care and anaesthesia, Ph D, Karolinska Institutet
Other Study IDs: Barotrauma COVID-19
Record Dates: First submitted 2023-05-25; First posted 2023-05-26 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Barotrauma
MeSH Terms: conditions — COVID-19; Barotrauma | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Respiratory support by an open system
  Interventions: Procedure: Open system
- Respiratory support by non-invasive mechanical ventilation
  Interventions: Procedure: Non-invasive mechanical ventilation
- Respiratory support by invasive mechanical ventilation
  Interventions: Procedure: Invasive mechanical ventilation

INTERVENTIONS:
Procedure: Open system — Oxygen delivered on open system, for example high flow nasal cannula or low flow oxygen by nasal cannula or face mask
  Groups: Respiratory support by an open system
Procedure: Non-invasive mechanical ventilation — Respiratory support by for example continues or bilevel positive airway pressure
  Groups: Respiratory support by non-invasive mechanical ventilation
Procedure: Invasive mechanical ventilation — Respiratory support delivered through endotracheal tube or tracheostomy
  Groups: Respiratory support by invasive mechanical ventilation

SUMMARY:
During the pandemic of COVID-19, studies reporting a high incidence of barotrauma, both pneumothorax but also pneumomediastinum, in patients with critical COVID-19. If this is complications of the respiratory support used to treat patients hypoxemia or if it is a direct consequence of COVID-19 damaging the lung tissue is not known.

The aim of this study is to investigate the incidence and type barotrauma, if there is an association between barotrauma and level of respiratory support used in the intensive care unit, and if barotrauma is associated with worse outcome compared to patients without barotrauma.

ELIGIBILITY:
Inclusion Criteria:

* Positive polymerase chain reaction for SARS-CoV-2
* Admitted to ICU due to respiratory failure

Exclusion Criteria:

* Transferred to or from an ICU in other hospital/region making data collection regarding baseline data/outcomes not possible

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with critical COVID-19 admitted to an intensive care unit at Södersjukhuset, Stockholm, Sweden, March 2020 to May 2021.
Sampling Method: Probability Sample
Enrollment: 669 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Barotrauma | 28 days from ICU admission
  Pneumothorax, pneumomediastinum, pneumatocele or subcutaneous emphysema as verified by radiology

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Jonmarker, Ph D, Principal Investigator — Stockholm South General Hospital
Locations (1):
- Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participants data for our patients is protected by law and can therefore not be made available for other researchers.

REFERENCES:
- [Derived] Jensen AL, Litorell J, Grip J, Dahlberg M, Joelsson-Alm E, Jonmarker S. A descriptive, retrospective single-centre study of air-leak syndrome in intensive care unit patients with COVID-19. Acta Anaesthesiol Scand. 2025 Mar;69(3):e14582. doi: 10.1111/aas.14582. PMID 39936659